CLINICAL TRIAL: NCT05613023
Title: PACE-NODES. A Phase III Randomised Trial of 5 Fraction Prostate SBRT Versus 5 Fraction Prostate and Pelvic Nodal SBRT
Brief Title: A Trial of 5 Fraction Prostate SBRT Versus 5 Fraction Prostate and Pelvic Nodal SBRT
Acronym: PACE-NODES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Prostate Cancer UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR5545; Prostate Cancer UK (Other Grant/Funding Number: MA-CT20-005)
Record Dates: First submitted 2022-03-07; First posted 2022-11-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-SBRT (Active Comparator): Participants allocated P-SBRT will receive 36.25Gy in 5 fractions to the prostate and seminal vesicles on alternate days (40Gy to prostate CTV).
  Interventions: Radiation: SBRT
- PPN-SBRT (Experimental): Participants allocated PPN-SBRT will receive 36.25Gy in 5 fractions to the prostate and seminal vesicles on alternate days (40Gy to prostate clinical target volume (CTV)) and 25Gy in 5 fractions to pelvic nodes on alternate days.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiotherapy
  Other Names: SABR

SUMMARY:
This study will compare the safety and efficacy of curative radiotherapy to the prostate and lymph glands given in 5 visits to that of prostate alone radiotherapy given in 5 visits, in men with high risk localised prostate cancer.

DETAILED DESCRIPTION:
This study will look at the safety of curative radiotherapy to the prostate and lymph glands given in 5 visits, in men with high risk localised prostate cancer.

The purpose of the research is to test an advanced type of external beam radiotherapy called stereotactic body radiotherapy (also known as SBRT) in 1128 participants with high risk localised prostate cancer (that is, prostate cancer that has not spread beyond the prostate gland but is at high risk of growing quickly or spreading). Importantly, this treatment delivers a potentially curative dose of radiotherapy in only 5 treatments over two weeks. Half the participants in the trial will receive radiotherapy to the prostate, the other half will have radiotherapy to the prostate as well as the surrounding lymph nodes. The investigators will follow patients in the trial for at least three and half years to see which treatment is best. The investigators will be looking at whether it is safe to give this treatment by reviewing any side-effects that occur and also assessing whether giving SBRT to the lymph nodes as well as the prostate reduces the chance of prostate cancer returning.

The treatment will take place at NHS radiotherapy centres that are experienced in giving SBRT and radiotherapy to the pelvic nodes, and have been quality assured to deliver these treatments

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at randomisation
2. Histopathological confirmation of prostate adenocarcinoma with Gleason/ISUP grade group scoring within twelve months of randomisation (unless otherwise discussed with the CI or co-Clinical Leads)
3. Patients planned for 12-36 months androgen deprivation therapy
4. High risk localised prostate cancer as defined by

   * Gleason 8-10 (grade groups 4 and 5) and/or
   * Stage T3a/b or T4 and/or
   * PSA > 20ng/ml (or >10 ng/ml for patients on 5-alpha reductase inhibitors)
5. Multi-parametric MRI of the pelvis- to include at least one functional MRI sequence in addition to T2W imaging within twelve months of randomisation
6. Radiological staging to exclude metastatic disease, prior to starting ADT, with one of the following: PSMA PET-CT, fluciclovine/choline PET-CT, whole-body MRI, bone scan, CT of chest, abdomen and pelvis (imaging method as per local practice/standard of care).
7. WHO performance status 0-2
8. Ability of research subject to give written informed consent

Exclusion Criteria:

1. N1 or M1 disease
2. PSA >50ng/ml (or >25ng/ml for patients on 5-alpha reductase inhibitors), unless PET-CT imaging has been performed to confirm N0M0 disease
3. Previous active treatment for prostate cancer
4. Patients where SBRT is contraindicated: prior pelvic radiotherapy, inflammatory bowel disease, significant lower urinary tract symptoms N.B. where patient has repeated imaging showing bowel in close apposition to target volumes that would make pelvic radiotherapy highly unlikely to be deliverable should be excluded.
5. Contraindications to fiducial marker insertion, where used- including clotting disorders, or patients at high risk when stopping anticoagulation or antiplatelet medications
6. Bilateral hip prostheses or any other implants/hardware that would introduce substantial CT artefacts and would make pelvic node planning more difficult.
7. Patients who have had chemotherapy within 6 weeks of the start of radiotherapy.
8. Life expectancy < 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Time to biochemical or clinical failure | minimum of 3.5 years follow up post-randomisation
  Time to biochemical or clinical failure as defined by time from randomisation to the first progression event (either biochemical failure, local recurrence, lymph node/pelvic recurrence, distant metastases, recommencement of androgen deprivation therapy or death due to prostate cancer).

SECONDARY OUTCOMES:
Clinical reported acute toxicity | 12 weeks post-randomisation
  Clinical reported acute and late toxicity using CTCAE version 5.0 and RTOG criteria. Focus will be given to GU and GI Grade 2 or higher (G2+) toxicities
Clinical reported late toxicity | up to 5 years post-randomisation
  Clinical reported acute and late toxicity using CTCAE version 5.0 and RTOG criteria. Focus will be given to GU and GI Grade 2 or higher (G2+) toxicities
Metastatic relapse-free survival | up to 5 years post-randomisation
  Time from randomisation to distant metastases or death from prostate cancer
Prostate cancer-specific survival | up to 5 years post-randomisation
  Time from randomisation to death due to prostate cancer
Overall survival | up to 5 years post-randomisation
  Time from randomisation to death from any cause
Patient Reported Outcome Measures | up to 5 years post-randomisation
  Quality of life will be evaluated using combined data from the following questionnaires. IPSS questionnaire: a validated diagnostic tool used to assess urinary & bowel incontinence.
  IIEF-5: validated diagnostic tool for erectile dysfunction. EPIC questionnaire: to assess typical symptoms after radiotherapy in prostate cancer patients. EQ-5D: a commonly used generic questionnaire to measure health-related QoL used to asess mobility, self-care, usual activities, pain/discomfort, anxiety/depression & the subject's perceptions of their own current overall health. A QoL analysis plan will be developed in consultation with the TMG with key endpoints for each questionnaire. Standard algorithms will be used to derive scores and handle missing data. Changes from baseline at each time point will be compared within groups as well as between treatment groups (by means of ordinal logistic regressions or ANCOVA models). Analyses to account for the longitudinal nature of the data may be used.
Adherence to radiotherapy protocol | after completion of treatment
  Qualitative analysis of adherence to pre-specified radiotherapy dose constraints with radiotherapy quality assurance to demonstrate feasibility in a muliticentre setting.

CONTACTS AND LOCATIONS:
Locations (42):
- Ireland (3):
  - Bon Secours Radiotherapy Cork in partnership with UPMC Hillman Cancer Centre, Cork
  - St Lukes Radiation Oncology Network, Dublin
  - Mid Western Radiation Oncology Centre, Limerick
- Auckland Hospital, Auckland, New Zealand
- United Kingdom (38):
  - James Cook University Hospital, Middlesbrough, South Tees
  - Worcestershire Acute Hospitals Nhs Trust, Worcester, Worcestershire
  - Belfast City Hospital, Belfast
  - Bristol Haematology and Oncology Centre, Bristol
  - West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - University Hospitals of Derby & Burton NHS Foundation Trust, Derby
  - North Middlesex University Hospital NHS Trust, Edmonton
  - Royal Devon & Exeter, Exeter
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Mount Vernon Cancer Centre, Hillingdon
  - East Suffolk & North Essex NHS Foundation Trust, Ipswich
  - Queen Elizabeth Hospital, Kings Lynn
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - United Linconshire Hospitals NHS Trust, Lincoln
  - Guy's and St Thomas' Hospital NHS Foundation Trust, London
  - Royal Free Hospital, London
  - St Bartholomew's Hospital, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle upon Tyne
  - Northampton General Hospital NHS Trust, Northampton
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospital NHS Trust, Nottingham
  - Churchill Hospital, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Portsmouth Hospitals University NHS Trust, Portsmouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Mid and South Essex NHS Foundation Trust, Southend
  - University Hospital North Midlands NHS Trust, Stoke-on-Trent
  - Royal Marsden Hospital, Sutton
  - Torbay and South Devon NHS Foundation Trust, Torquay
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Undecided